CLINICAL TRIAL: NCT02495818
Title: Suprascapular Nerve Block Guided by Ultrasound in the Rehabilitation of the Supraspinatus Tendonitis - A Randomized Double Blind Controlled Trial
Brief Title: Suprascapular Nerve Block Guided by Ultrasound
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marta Imamura (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, Coordinator of the Clinical Research Center for Physical and Rehabilitation Medicine of HC FMUSP, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Suprascapular Nerve Block
Record Dates: First submitted 2015-07-01; First posted 2015-07-13 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Rotator Cuff Syndrome
Keywords: Rotator cuff syndrome; supraspinatus tendonitis; suprascapular nerve block; ultrasound guided; supraspinatus
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Suprascapular nerve block with infusion of 5ml lidocaine at 2%, guided by Ultrasound combined with homemade exercises (Codman and Hughston exercises).
  Interventions: Procedure: Lidocaine; Other: Homemade exercises
- Saline solution (Sham Comparator): Intervention with suprascapular nerve block with 5ml saline solution guided by Ultrasound combined with homemade exercises (Codman and Hughston exercises).
  Interventions: Procedure: Saline solution; Other: Homemade exercises

INTERVENTIONS:
Procedure: Lidocaine — Suprascapular Nerve Block Guided by Ultrasound with 5ml lidocaine at 2%.
  Arms: Lidocaine
Procedure: Saline solution — Suprascapular Nerve Block Guided by Ultrasound with 5ml saline solution
  Arms: Saline solution
Other: Homemade exercises — Codman and Hughston exercises.

SUMMARY:
The purpose of this study is to evaluate the effect of suprascapular nerve block guided by ultrasound combined with home exercises compared with placebo. Pain intensity, function, pressure pain threshold and goniometry were designed to be assessed in all patients.

DETAILED DESCRIPTION:
The trial is being carried out in the Institute of Physical Medicine and Rehabilitation of the University of São Paulo since June 2013. The investigators are including patients with clinical diagnosis of supraspinatus tendinitis based on the Lateral Jobe Test.

The patients are being randomized in two arms: Active (2% 5ml lidocaine for suprascapular nerve block and home exercises) and placebo control (saline solution as the nerve block and home exercises). The randomization is being performed in blocks of 4 and 6.

The investigator, the raters, the MD who makes the procedure and the patients are blind to treatment.

4 visits are being performed. Screening and initial evaluation visit, procedure visit, follow up 1 week after intervention and follow up 12 weeks after intervention.

The sample size was estimated to be 54 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of supraspinatus tendonitis, based on Jobe's lateral test;
* Pain longer than 1 month prior to screening visit;
* BMI between 20 and 30 kg/m²;
* VAS of 4 or higher in screening visit;
* Ability to understand the questionaires and instructions for home exercises;
* Signed Informed Consent Form;

Exclusion Criteria:

* History of:

  1. Shoulder surgery;
  2. Athletic activities;
  3. Severe shoulder arthrosis;
  4. Diagnosis of total rupture of supraspinatus tendon
  5. Autoimmune disease;
  6. Fracture of humerus, acromion and clavicle
  7. Luxation and subluxation of shoulder.
  8. Diseases that cause spasticity, such as stroke or spinal cord injury;
  9. Systemic alterations that can lead to peripheral neuropathy;
  10. Uncontrolled Diabetes or thyroidopathy;
  11. Diagnosis of cervical spinal cord injury that results in motor alterations;
  12. Allergy or hypersensibility for local or systemic anaesthetics;
  13. Coagulopathy;
  14. Fibromyalgia according to the 1990 American School of Rheumatology;
  15. Uncontrolled psychiatric diseases or controlled psychiatric diseases that need more than two medicines;
  16. Acute of chronic renal failure;
  17. Pulmonary diseases that presents hypoxemia such as Gold IV Chronic Obstructive Pulmonary Disease or pulmonary fibrosis.
  18. Arrhythmia (except isolated supraventricular extrasystoles), coronary failure or functional class 2 or higher heart failure
* Pregnancy;
* Use of oral or subcutaneous anticoagulation agent;
* Patients who fail to comply with the proposed treatment.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the score of pain and function as assessed by Shoulder Pain and Disability Index (SPADI) | Baseline and one week after intervention
  Scale for assessing pain and shoulder function.

SECONDARY OUTCOMES:
Change from baseline in pain Intensity assessed by Visual Analogue Scale (VAS). | Baseline and one week after intervention.
  Self rated pain scale from 0 (no pain) to 10 (the maximum possible pain)
Change from baseline in pain Intensity assessed by Visual Analogue Scale (VAS). | Baseline and twelve weeks after intervention.
  Self rated pain scale from 0 (no pain) to 10 (the maximum possible pain)
Change from baseline in the score of pain and function as assessed by SPADI | Baseline and 12 weeks after intervention
  Scale for assessing pain and shoulder function.
Change from baseline in Pain Pressure Threshold (PPT) as assessed by Algometry | Baseline and one week after intervention
  Measurement of pain under pressure of the structures of dermatome, myotome and sclerotome corresponding to levels C5 and C6 of spinal cord.
Change from baseline in Pain Pressure Threshold (PPT) as assessed by Algometry | Baseline and twelve weeks after intervention
  Measurement of pain under pressure of the structures of dermatome, myotome and sclerotome corresponding to levels C5 and C6 of spinal cord.
Change from baseline in Active Range of Motion (AROM) as assessed by Goniometry | Baseline and one week after intervention
  Goniometry for active movements for flexion and abduction of the shoulder
Change from baseline in Active Range of Motion (AROM) as assessed by Goniometry | Baseline and twelve weeks after intervention
  Goniometry for active movements for flexion and abduction of the shoulder
Safety as assessed by the number of Adverse Events | 1 week and 12 weeks after intervention
  Assessment of possible Adverse Events after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otani PT, Rached RDVA, Alfieri FM, de Azevedo Neto RS, Hsing WT, Battistella LR, Imamura M. Ultrasound-guided suprascapular nerve block with lidocaine vs. saline combined with physical exercises for the rehabilitation of supraspinatus tendinitis: a randomized double-blind controlled trial. Front Pain Res (Lausanne). 2024 Nov 12;5:1490320. doi: 10.3389/fpain.2024.1490320. eCollection 2024. PMID 39600565